CLINICAL TRIAL: NCT02653677
Title: Glycemic and Hormone Responses and Satiety After the Intake of Four Types of Bread.
Brief Title: Glycemic and Hormone Responses After the Intake of Four Types of Bread.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Simona Bo, MD, University of Turin, Italy
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Bo11/14
Record Dates: First submitted 2016-01-06; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Hyperglycemia; Insulin Sensitivity
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- commercial bread, wheat flour (Active Comparator): Intake of the specific kind of bread
  Interventions: Other: intake of the specific kind of bread
- wheat, organic flour (Experimental): Intake of the specific kind of bread
  Interventions: Other: intake of the specific kind of bread
- wheat, supermarket flour (Experimental): Intake of the specific kind of bread
  Interventions: Other: intake of the specific kind of bread
- einkorn, organic flour (Experimental): intake of the specific kind of bread
  Interventions: Other: intake of the specific kind of bread

INTERVENTIONS:
Other: intake of the specific kind of bread — To determine the glycemic and insulinemic responses (area-under the curve, AUCs), the satiety rate and the AUCs of free fatty acids (FFA), triglycerides and ghrelin after the ingestion of four types of breads, each containing 50g of available carbohydrates

SUMMARY:
The purposes of the present study are to determine the glycemic and insulinemic responses, the satiety rate and the postprandial plasma concentrations of free fatty acids, triglycerides and satiety hormones after the ingestion of four types of breads: handcrafted bread made with wheat organic flour; handcrafted bread with wheat flour of large-scale retail distribution; handcrafted bread with organic einkorn flour and a commercial wheat bread.

DETAILED DESCRIPTION:
The postprandial blood glucose concentration appears to play a critical role in the development of diabetes and cardiovascular diseases; it is largely influenced by the carbohydrate load of a meal. Thus, advocating carbohydrate (CHO) foods that promote favorable glycemic and insulinemic responses, with maintenance of satiety high over a longer period, may be a beneficial approach against many chronic diseases.

Bread is a basic food in Italian feeding. The industrial production of bread is gradually replacing the craft production by small bakeries. It is possible to buy daily bread obtained by completing baking carried out directly at the point of sale from pre-cooked and frozen dough. The use of "improver" as enzyme preparations such as alpha-amylase, improves the quality of bread. A study has found that trestatin, an amylase inhibitor incorporated into bread, produced lower glycemic and insulinemic responses; another has reported that bread made from the ancient wheat Einkorn (Triticum monococcum) elicited a reduced production of glucose-dependent insulinotrophic polypeptide (GIP).

The objectives of the present study are to determine the glycemic and insulinemic responses (area-under the curve, AUCs), the satiety rate and the AUCs of free fatty acids (FFA), triglycerides and ghrelin after the ingestion of four types of breads, each containing 50g of available CHO:

* 97 g handcrafted bread made with wheat organic flour;
* 97 g handcrafted bread with wheat flour of large-scale retail distribution;
* 94 g handcrafted bread with organic einkorn flour
* 86 g commercial precooked-frozen white bread.

  16 healthy volunteers participated to this randomized cross-over trial. Each participant consumed the specific portion of a type of bread in the morning, after 8-12 h fasting. The other 3 types of bread are consumed by participants in the order determined by the randomization procedure, after a week each other.

At enrollment, all participants meet the inclusion criteria (see below). Nutrition and exercise advices are given for the day before each bread test. Participants should consume the bread portion in 15 minutes.

Blood samples are drawn every 30-min from fasting until 120-min after bread consumption. The following variables are evaluated at each time point: glucose, insulin, FFA, triglycerides, acylated ghrelin. The satiety rate is estimated every 30-min by the Satiety Labeled Intensity Magnitude scales.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 18 and 25 kg/m2
* healthy
* Accept to participate in the study

Exclusion Criteria:

* smokers
* subjects suffering from any diseases
* drug therapy
* dietary supplementation
* patients unable to give informed consent to participate in the study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Glucose-under-the curve (AUC) after ingestion of 4 types of bread | 0 to 120 minutes after the ingestion of each bread
  Glycemic AUC is defined as the blood glucose increment over 2 hours in response to the consumption of the amount of bread providing 50 g of available carbohydrates

SECONDARY OUTCOMES:
Insulin-under-the curve (AUC) after ingestion of 4 types of bread | 0 to 120 minutes after the ingestion of each bread
  Insulinemic AUC is defined as the blood insulin increment over 2 hours in response to the consumption of the amount of bread providing 50 g of available carbohydrates

OTHER OUTCOMES:
Free fatty acid (FFA) AUC after the ingestion of 4 types of bread | 0 to 120 minutes after the ingestion of each bread
  FFA AUC is defined as the variation in FFA concentrations in response to the consumption of the amount of bread providing 50 g of available carbohydrates
Ghrelin responses after the ingestion of 4 types of bread | 0 to 120 minutes after the ingestion of each bread
  Ghrelin AUC is defined as the variation in ghrelin concentrations in response to the consumption of the amount of bread providing 50 g of available carbohydrates

CONTACTS AND LOCATIONS:
Overall Officials: Simona Bo, MD, Principal Investigator — University of Turin, Italy